CLINICAL TRIAL: NCT06049251
Title: Effects of ELDOA Technique Versus Lumbar SNAGS With Motor Control Exercises on Pain, Function and Mobility in Patients With Chronic Low Back Pain.
Brief Title: ELDOA Technique Versus Lumbar SNAGS With Motor Control Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0131 Anam Hamid
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Low Back Pain
Keywords: Core stability; Disability; Low Back Pain; Stretching Exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELDOA exercises (Experimental): ELDOA exercises
  Interventions: Other: ELDOA exercises
- Lumbar SNAGS and motor control exercises (Active Comparator): Lumbar SNAGS and motor control exercises
  Interventions: Other: Lumbar SNAGS and motor control exercises

INTERVENTIONS:
Other: ELDOA exercises — The patients will be asked to sit down on a floor in upright position and keep their legs apart and knees semi-flexed, feet in outward and upward position, knees constantly pushing downwards, straight lower back, raise arms with palms facing upward, and chin should be pulled back.
  ELDOA stretch for L5-S1 level Patients will be asked to lay on floor and flatten and bring their legs up and straight with the support of wall, straight knees and keep distance between them, connect their toes, raise arm and externally rotate with wrist extension than press their heels and palms out.
  ELDOA exercises will be performed with 2 sets of 5 repetitions with 45 second hold and15 sec rest between each set once a day.
  Arms: ELDOA exercises
Other: Lumbar SNAGS and motor control exercises — The patient will be seated and his pelvis will be stabilized with belt at the level of the anterior superior iliac spine while the SNAGs are administered. The ulnar aspect of the therapist's hand will be placed over the spinous processes of the affected segment's superior vertebrae, for flexion glide and inferior vertebrae for extension glide respectively. A passive glide will be applied and kept up until the patient finished a full movement arc. The glides will be given for six repetitions for three sets every session. Glide can be given unilateral for other movements.
  Motor Control Exercises:
  Exercise training with 7sec Hold and 10 reps
  Arms: Lumbar SNAGS and motor control exercises

SUMMARY:
Study will be a Randomized clinical trial to check the effects of ELDOA technique versus lumbar SNAGS with motor control exercises on pain, function and mobility in patients with chronic low back pain. Duration of study will be 8 months, non probability convenience sampling technique will be used, subject following eligibility criteria from District Headquarters Hospital Okara will be randomly allocated in two groups using computer random number generator. baseline assessment will be done. Group A participants will be given baseline treatment along with ELDOA exercises, Group B participants will be given baseline treatment along with Lumbar SNAGS and motor control exercises for 3 weeks. Assessment will be done by using Numeric Pain Rating Scale, Oswestry Disability Index and Inclinometer at baseline, at 3 weeks and a follow up will be taken at 6 weeks. 3 sessions per week will be given, data will be analyzed by using SPSS version 21.

DETAILED DESCRIPTION:
LBP is a significant global health problem, and its impact is still great. In 2019, there were 6972.5 (95% UI 6190.5 to 7860.5) age-standardized point prevalence estimates for LBP worldwide, with 568.4 million (95% UI 505.0 to 640.6 million) prevalent cases. The GBD research also revealed that LBP has a worldwide point prevalence of 9.4%, with men having a greater prevalence than women (8.7% vs. 10.1%). Back discomfort might arise as a result of mobility disorders, musculoskeletal sprains, incorrect spine positioning, or nucleus pulposus degeneration. There is huge literature regarding the management of low back pain and yet after the decades of research there are gaps in treatment options. The current study will compare the ELDOA technique to Lumbar SNAGS with motor control exercises. The current study is novel in a way that there is very limited evidence avialbale on ELDOA Technique and Motor Control Exercises. This study will provide vital insights into their efficacy and can help to guide clinical decision making for individuals with low back pain. Furthermore, this study can add to the expanding body of information regarding low back pain treatment and will help to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30
* Patients of both genders.
* Patients having chronic Low Back Pain ( >3 months duration)
* Patients with restricted range of motion (patients will be examined for active lumbar range of motion)
* Patients with lumbar straightening based on referral from orthopedic

Exclusion Criteria:

* History of neurological condition of hip and lumbar region.
* Medical red flag history (tumor, metabolic diseases, rheumatoid arthritis, osteoporosis or Infection)
* Medical record of severe disabling chronic cardiovascular and pulmonary disease.
* Prescribed history of epidural steroidal injection for pain.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 3rd Week
  The 11-point NPRS (intervals from 0-10) is used to quantify pain intensity; 0 represents no pain, and 10 represent the worst possible agony
Oswestry Disability Index | 3rd Week
  Questionnaire examines perceived level of disability in 10 everyday activities of daily living. Test-retest reliability has been shown to be high, a study by Fairbank et al recorded values ranging from = 0.83 to 0.99 that can vary over a given period of time. Each item consists of 6 statements. With Each item is scored on a 0---5 scale, and the maximum score is 50.
Inclinometer | 3rd Week
  Lumbar spine mobility will be assessed by inclinometer. It consists of a circular, fluid- filled disk with a bubble that indicates the number of degrees on the scale of protractor.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Principal Investigator — Riphah International University, Lahore, pakistan
Locations (1):
- DHQ, Okāra, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen S, Chen M, Wu X, Lin S, Tao C, Cao H, Shao Z, Xiao G. Global, regional and national burden of low back pain 1990-2019: A systematic analysis of the Global Burden of Disease study 2019. J Orthop Translat. 2021 Sep 10;32:49-58. doi: 10.1016/j.jot.2021.07.005. eCollection 2022 Jan. PMID 34934626
- [Background] Ma K, Zhuang ZG, Wang L, Liu XG, Lu LJ, Yang XQ, Lu Y, Fu ZJ, Song T, Huang D, Liu H, Huang YQ, Peng BG, Liu YQ. The Chinese Association for the Study of Pain (CASP): Consensus on the Assessment and Management of Chronic Nonspecific Low Back Pain. Pain Res Manag. 2019 Aug 15;2019:8957847. doi: 10.1155/2019/8957847. eCollection 2019. PMID 31511784
- [Background] 3. Chitale N, Patil D, Phansopkar P. Efficacy of Integrated Neuromuscular Inhibition Technique Versus Mulligan Mobilization on Pain and Functional Disability in Subjects with Non-Specific Low Back Pain-A Research Protocol. Journal of Pharmaceutical Research International. 2021:99-104
- [Background] Shahzad M, Rafique N, Shakil-Ur-Rehman S, Ali Hussain S. Effects of ELDOA and post-facilitation stretching technique on pain and functional performance in patients with piriformis syndrome: A randomized controlled trial. J Back Musculoskelet Rehabil. 2020;33(6):983-988. doi: 10.3233/BMR-181290. PMID 32894238
- [Background] Stuge B. Evidence of stabilizing exercises for low back- and pelvic girdle pain - a critical review. Braz J Phys Ther. 2019 Mar-Apr;23(2):181-186. doi: 10.1016/j.bjpt.2018.11.006. Epub 2018 Nov 17. PMID 30471967
- [Background] 7. Salik S, Rani S, Hayat R, Manzoor S, Malik AU, Maqbool S. Comparison between Mulligan Sustained natural apophyseal glides (snags) VS McKenzie exercises in Chronic Mechanical Low back pain. Pakistan Journal of Medical & Health Sciences. 2022;16(10):141-.
- [Background] 8. Shamshad M, Kanwal R, Butt R, Haider HMM. Effects of ELDOA technique versus McKenzie extension exercises on non-specific low back pain patients.: a randomized clinical trial. The Rehabilitation Journal. 2022;6(03):429-34.
- [Background] Bhat P V, Patel VD, Eapen C, Shenoy M, Milanese S. Myofascial release versus Mulligan sustained natural apophyseal glides' immediate and short-term effects on pain, function, and mobility in non-specific low back pain. PeerJ. 2021 Mar 15;9:e10706. doi: 10.7717/peerj.10706. eCollection 2021. PMID 33777508
- [Background] Ibrahim AA, Akindele MO, Ganiyu SO. Effectiveness of patient education plus motor control exercise versus patient education alone versus motor control exercise alone for rural community-dwelling adults with chronic low back pain: a randomised clinical trial. BMC Musculoskelet Disord. 2023 Feb 23;24(1):142. doi: 10.1186/s12891-022-06108-9. PMID 36823567